CLINICAL TRIAL: NCT06461754
Title: Prediction of Successful Liberation From Invasive Mechanical Ventilation Via Lung and Diaphragmatic Ultrasound in Intensive Care Unit Patients, Prospective, Observational Study
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fawzy Abbas Badawy, Assistant lecturer of anesthesia,intensive care and pain management sohag faculty of medicine, Sohag University
Other Study IDs: Soh-Med-22-09-20
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Liberation From Mechanical Ventilation in ICU Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (2):
- Succeeded Group (SG): Group of patients who succeeded weaning from mechanical ventilation
  Interventions: Other: Sonographic evaluation of diaphragm and lung
- Failed Group (FG): Group of patients who failed weaning from mechanical ventilation
  Interventions: Other: Sonographic evaluation of diaphragm and lung

INTERVENTIONS:
Other: Sonographic evaluation of diaphragm and lung — While the patient in a semi-sitting position (20-40 degree), by ultrasound, the diaphragm thickness was measured in the zone of apposition, on the mid-axillary line among the 8th and 10th intercostal spaces, using a 7-10 MHz linear probe in (M) mode. at the end of expiration and at the end of inspiration by capturing nearly three images during spontaneous patient breathing. The average of three DTI measurements was calculated In lung ultrasound, 2-4 MHz convex ultrasound probe in (B) mode was employed. We implemented a modified LUSm in our investigation, which assessed four lung regions on each side.

SUMMARY:
Liberation from invasive mechanical ventilation (IMV) remains a challenge for intensive care physicians. Although standard indices such as blood gases and respiratory clinical data are used routinely but they still have some limitations. Diaphragmatic and lung sonographic parameters (pulmonary scores) recently became the hot spot to help in anticipation of liberation from IMV.The aim of this study was to ensure that, sonographic diaphragmatic thickening indices and lung scores are reliable and accurate additional tools to anticipate successful liberation from IMV in intensive care unit (ICU) patients.

Methods: This study was a prospective, observational study conducted at Sohag university hospital on 80 patients admitted to the Intensive Care Unit (ICU) and mechanically ventilated invasively for more than 24 hours and they were ready for weaning by standard methods. At the time of spontaneous breathing trials (SBT), we did diaphragm and lung ultrasound, where we applied diaphragmatic thickening indices (DTI) and a modified lung ultrasound scores (LUSm). Patients classified into two groups; failed group (FG) and (SG) of liberation from IMV. Comparison between (FG) and (SG) in relation to pulmonary scores (DTI and LUSm) were recorded. Cut-off values, sensitivity and specificity for DTI and LUSm were obtained. Also, comparison between (FG) and (SG) in relation to demographic, clinical and respiratory data were assessed and all data were statistically analysed.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age, more than 24 hours on IMV, and prepared for weaning

Exclusion Criteria:

* A spinal cord injury that exceeded T8, arrhythmias, heart failure, hemodynamic instability, terminal extubation, pregnancy, pneumothorax, pneumomediastinum, COPD, thoracostomy, chest injuries that impeded ultrasound, pleural lesions, or neuromuscular diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 80 patients who were admitted to the ICU and on invasive mechanical ventilation for more than 24 hours and ready for weaning
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
a cut off values for DTI and LUSm with sensitivity and specificity for anticipation of liberation from invasive mechanical ventilation | One year
  we reporte a cut-off value for DTI and LUSm below or above which the risk for failure of weaning can be predicted with a sensitivity persent and a specificity persent.

SECONDARY OUTCOMES:
The correlations of DTI and LUSm with demographic, clinical and respiratory data | one year
  We recorded the relations of DTI and LUSm with demographic, clinical and respiratory data in prediction of succeeded liberation from IMV

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol

REFERENCES:
- [Background] Tenza-Lozano E, Llamas-Alvarez A, Jaimez-Navarro E, Fernandez-Sanchez J. Lung and diaphragm ultrasound as predictors of success in weaning from mechanical ventilation. Crit Ultrasound J. 2018 Jun 18;10(1):12. doi: 10.1186/s13089-018-0094-3. PMID 29911284
- [Background] Gok F, Mercan A, Kilicaslan A, Sarkilar G, Yosunkaya A. Diaphragm and Lung Ultrasonography During Weaning From Mechanical Ventilation in Critically Ill Patients. Cureus. 2021 May 16;13(5):e15057. doi: 10.7759/cureus.15057. PMID 34007779
- [Background] Farghaly S, Hasan AA. Diaphragm ultrasound as a new method to predict extubation outcome in mechanically ventilated patients. Aust Crit Care. 2017 Jan;30(1):37-43. doi: 10.1016/j.aucc.2016.03.004. Epub 2016 Apr 22. PMID 27112953
- [Background] Ferrari G, De Filippi G, Elia F, Panero F, Volpicelli G, Apra F. Diaphragm ultrasound as a new index of discontinuation from mechanical ventilation. Crit Ultrasound J. 2014 Jun 7;6(1):8. doi: 10.1186/2036-7902-6-8. eCollection 2014. PMID 24949192